CLINICAL TRIAL: NCT05425043
Title: The Use of Granulocyte Transfusions After Umbilical Cord Blood Transplant for Leukaemia: a Prospective, Non-randomised, Single-centre Study to Evaluate Safety and Immune Reconstitution
Brief Title: Granulocyte Transfusions After Umbilical Cord Blood Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Children's Cancer and Leukaemia Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 295998
Record Dates: First submitted 2021-12-17; First posted 2022-06-21 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Cancer
Keywords: Granulocytes; HSCT; Haematopoietic Stem Cell Transplant; Pediatric; Leukemia
MeSH Terms: conditions — Neoplasms; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Granulocytes (Experimental): Patient to receive pooled granulocytes for 7 days concurrently. 20 participants will be approached for this arm.
  Interventions: Biological: Granulocytes
- Control (No Intervention): Non-randomised control arm, where patients who are receiving a stem cell transplant, as described in the eligibility criteria, are asked for a blood sample. This is to establish a baseline versus the experimental arm. 20 participants will be approached for this arm.

INTERVENTIONS:
Biological: Granulocytes — Receive granulocytes for 7 consecutive days after engraftment post transplant
  Arms: Granulocytes

SUMMARY:
Although most children with leukaemia are cured using drugs (chemotherapy) alone, for some children additional treatments are needed. Stem cell transplant can cure children where chemotherapy and other drugs have failed. In this case, the immune cells of the donor attack the leukaemia cells of the patient. Cord blood collected from the placenta of unrelated babies is often used as a donor cell source and appears to work well at controlling leukaemia and less likely to cause complications such as when the immune cells also mistakenly attack healthy tissues (called graft versus host disease, GVHD).

The investigators have noticed that during cord blood transplant, the donor immune system appears to recover more quickly and not be associated with GVHD, when a type of blood transfusion containing white cells are also given to the patient. The infused white cells appear to stimulate the donor immune cells to expand much more than usually seen.

During this research, the investigators will study this immune cell expansion during cord blood transplant in children with difficult-to-cure leukaemia who also receive a transfusion of white cells, termed granulocytes. The investigators will assess the safety of the effects of the white cell transfusions and the immune cell expansion on the child, and look at the outcomes on the patient's leukaemia, and whether there is GVHD or not.

DETAILED DESCRIPTION:
Most children with acute leukaemia are cured with chemotherapy alone but a few children are either refractory to such therapy, or relapse after it has been administered.

Some of these relapsed or refractory children are given HCT (hematopoietic cell transplantation), and some will be cured with HCT. HCT acts to cure children with leukaemia in two ways:

* There is chemotherapy given before the transplant, to get rid of recipient marrow and the recipient immune system. This chemotherapy is of higher dose than is given in standard chemotherapy protocols, and this dose escalation might overcome the resistance to chemotherapy that is inherent in children with relapsed or refractory disease.
* The engrafting immune system - derived from the HCT donor - recognises the residual leukaemia and rejects it. This is known as graft-versus-leukaemia, and this Is the main way that transplant cures refractory diseases.

Most children with refractory and / or relapsed leukaemia will die of their leukaemia. Transplant offers a chance of cure where conventional therapies will fail. Transplant works through this graft-versus leukaemia effect. This is related to graft-versus-disease (GVHD) and involves a recognition by donor derived T-cells of differences in the host leukaemia cells, and more generally in the recipient.

In general, the risk of relapse after transplant is:

* Reduced where there is graft versus host disease
* Reduced where the T-cells are left in the graft, a T-cell replete transplant. Often T-cells are removed from the graft - bone marrow, blood, or cord blood - to reduce the risk of GVHD
* Reduced where there is mismatch between the donor and recipient. The investigators and others have shown that it is possible to do T-cell replete, mismatched unrelated donor transplant in umbilical cord transplant.
* The risk of relapse is less in cord blood transplant compared to other cell sources, and this is particularly evident where there is residual disease present, and the risk of treatment failure is highest.
* The risk of chronic GVHD is reduced after cord blood transplant, even where the transplant is T-cell replete and there is mismatch between donor and recipient. Using adult donor-derived, mismatched donor transplant in a T-cell replete setting is associated with a risk of severe acute GVHD and chronic, extensive GVHD which limits quality of life.
* The most meaningful endpoint for children undergoing transplantation for any indication is disease-free and chronic GVHD-free survival. In malignancy this is best achieved using cord blood in a T-cell replete setting.

One of the investigators groups have published data from a xenograft model demonstrating that cord blood T-cells are better at controlling a human leukaemia than adult T-cells, and that the actual cord T-cells infiltrating the xenografted tumour are Cluster of Differentiation 810 (CD810). However, after T-cell replete transplant most of the recovering T-cells are Cluster of Differentiation 4 (CD4) and not Cluster of Differentiation (CD812). Childhood leukaemia is a rapidly proliferative disease, and experience tells us that relapse can happen early, within the first weeks and months. A graft versus tumour effect must be established quickly therefore, to prevent disease recurrence, and death from disease.

In this research, the investigators seek to replicate results that have been described and published prior. Here the investigators demonstrated early, transient, massive Cluster of Differentiation (CD8) T-cell reconstitution after cord blood transplantation without any chronic GVHD, despite early cessation of post-transplant immune suppression.

This observation is important since it incorporates the important components of a clinically meaningful graft-versus-leukaemia, from previous work:

* CD8 biased
* Cord blood
* T-cell replete setting
* Mismatched donors
* No chronic GVHD

This has been recognized by leaders in the field, and as part of the peer review of this work. Milano, an expert in Cord Blood transplant in refractory leukaemia has written that "this is not only economically beneficial but may also result in a paradigm shift for the treatment of patients with high-risk leukaemia's. "

The trial is funded by bone marrow transplant local funds and by funds generated specifically for this research by families, including families with difficult-to-cure, including multiple relapsed and refractory leukaemia. The rationale and patient summaries have been shared with those families, in support of their fundraising efforts. Families of children with such leukaemia understand how transplant works, the risk it generates and the implications when cell therapies also fail where conventional therapy has already failed. They are the best placed of all of us to understand this balance of risk of therapy with risk of treatment failure, and the best placed therefore to understand the rationale and scope of this research.

It is important to replicate the data that the investigators have published. It is important that in a trial setting that the investigators better define the safety of the immune cell expansion, and the nature of the T-cells that are derived. It is important research, for the reasons explained above, and recognised by Milano and other commentators.

There is a control group for T-cell expansion numbers, and for safety evaluations including cytokine release syndrome and engraftment kinetics. This is not an efficacy trial, and the relapsed, refractory leukaemia is rare in children, and so randomisation is not appropriate. The granulocyte doses are standard for children, and what the investigators reported in their preliminary experience.

ELIGIBILITY:
Inclusion Criteria:

1. Children, aged <16 years, undergoing a first allogeneic, unrelated donor, T-cell replete, umbilical cord blood HSCT for high risk acute leukaemia.
2. Availability of at least a 6/8 allelic matched cord blood, of adequate cell dose, after allele-level matching at HLA (Human Leukocyte Antigen)-A, -B, -C, and -DRB1
3. Informed consent by parent or guardian. Age appropriate Assent will also be collected in those Children age 16 and under.

Exclusion Criteria:

1. Patients participating in other HSCT clinical trial
2. The transplant not indicated according to National Health Service England (NHSE) and British Society of Bone Marrow Transplant (BSBMT) Paediatric Transplant Group.
3. Pooled Granulocyte Transfusion contraindicated for any reason
4. Previous T cell replete unrelated donor cord blood transplant
5. Patients with a previous history of sensitivity to granulocyte transfusion will be excluded from the study

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
What is the number of patients with grade 1-4 cytokine release syndrome, related to the granulocytes infusions? | 2 years
  This is to access safety of the granulocyte infusions.
What is the number of patients with allo-immunisation after the granulocyte infusions? | 2 years
  This is to access safety of the granulocyte infusions.

SECONDARY OUTCOMES:
What is the median day to neutrophil and to platelet engraftment, and compared with a control group of cord blood transplant recipients not receiving granulocytes? | 2 years
  This is to measure the effect that the granulocyte infusion course have on engraftment and on the disease
How many patients experience grade II-IV GvHD? | 2 years
  This is to measure the effect that the granulocyte infusion course have on engraftment and on the disease
What is the median disease-free and overall survival in this patient cohort? | 2 years
  This is to measure the effect that the granulocyte infusion course have on engraftment and on the disease
How many patients enter flow and molecular remission after the transplant? | 2 years
  This is to measure the effect that the granulocyte infusion course have on engraftment and on the disease
What is the median date of cessation of immune suppression after the transplant, and compared with a control group of cord blood transplant recipients not receiving granulocytes? | 2 years
  This is to measure the effect that the granulocyte infusion course have on engraftment and on the disease

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wynn, MD FRCPath, Study Chair — Royal Manchester Children's Hospital
Locations (1):
- Royal Manchester Childrens Hospital, MFT, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keating AK, Langenhorst J, Wagner JE, et al. The influence of stem cell source on transplant outcomes for pediatric patients with acute myeloid leukemia. Blood Adv. 2019;3(7):1118-1128. Blood Adv. 2020 Mar 24;4(6):1081. doi: 10.1182/bloodadvances.2020001753. No abstract available. PMID 32196555
- [Background] Deambrosis D, Lum SH, Hum RM, Poulton K, Ogden W, Jones S, Stanworth S, Bonney D, Hiwarkar P, Wynn RF. Immune cytopenia post-cord transplant in Hurler syndrome is a forme fruste of graft rejection. Blood Adv. 2019 Feb 26;3(4):570-574. doi: 10.1182/bloodadvances.2018026963. PMID 30787020
- [Background] Lum SH, Miller WP, Jones S, Poulton K, Ogden W, Lee H, Logan A, Bonney D, Lund TC, Orchard PJ, Wynn RF. Changes in the incidence, patterns and outcomes of graft failure following hematopoietic stem cell transplantation for Hurler syndrome. Bone Marrow Transplant. 2017 Jun;52(6):846-853. doi: 10.1038/bmt.2017.5. Epub 2017 Feb 20. PMID 28218755
- [Background] Eapen M, Wang T, Veys PA, Boelens JJ, St Martin A, Spellman S, Bonfim CS, Brady C, Cant AJ, Dalle JH, Davies SM, Freeman J, Hsu KC, Fleischhauer K, Kenzey C, Kurtzberg J, Michel G, Orchard PJ, Paviglianiti A, Rocha V, Veneris MR, Volt F, Wynn R, Lee SJ, Horowitz MM, Gluckman E, Ruggeri A. Allele-level HLA matching for umbilical cord blood transplantation for non-malignant diseases in children: a retrospective analysis. Lancet Haematol. 2017 Jul;4(7):e325-e333. doi: 10.1016/S2352-3026(17)30104-7. Epub 2017 Jun 13. PMID 28623181
- [Background] Veys P, Danby R, Vora A, Slatter M, Wynn R, Lawson S, Steward C, Gibson B, Potter M, de la Fuente J, Shenton G, Cornish J, Gennery A, Snowden JA, Bonney D, Velangi M, Ruggeri A, Gluckman E, Hough R, Rocha V; British Society of Blood and Marrow Transplantation and Eurocord. UK experience of unrelated cord blood transplantation in paediatric patients. Br J Haematol. 2016 Feb;172(3):482-6. doi: 10.1111/bjh.13914. Epub 2016 Jan 5. No abstract available. PMID 26728432
- [Background] Boelens JJ, Aldenhoven M, Purtill D, Ruggeri A, Defor T, Wynn R, Wraith E, Cavazzana-Calvo M, Rovelli A, Fischer A, Tolar J, Prasad VK, Escolar M, Gluckman E, O'Meara A, Orchard PJ, Veys P, Eapen M, Kurtzberg J, Rocha V; Eurocord; Inborn Errors Working Party of European Blood and Marrow Transplant group; Duke University Blood and Marrow Transplantation Program; Centre for International Blood and Marrow Research. Outcomes of transplantation using various hematopoietic cell sources in children with Hurler syndrome after myeloablative conditioning. Blood. 2013 May 9;121(19):3981-7. doi: 10.1182/blood-2012-09-455238. Epub 2013 Mar 14. PMID 23493783
- [Background] Aldenhoven M, Jones SA, Bonney D, Borrill RE, Coussons M, Mercer J, Bierings MB, Versluys B, van Hasselt PM, Wijburg FA, van der Ploeg AT, Wynn RF, Boelens JJ. Hematopoietic cell transplantation for mucopolysaccharidosis patients is safe and effective: results after implementation of international guidelines. Biol Blood Marrow Transplant. 2015 Jun;21(6):1106-9. doi: 10.1016/j.bbmt.2015.02.011. Epub 2015 Feb 20. PMID 25708213
- [Background] Takami A. Hematopoietic stem cell transplantation for acute myeloid leukemia. Int J Hematol. 2018 May;107(5):513-518. doi: 10.1007/s12185-018-2412-8. Epub 2018 Jan 27. PMID 29374826
- [Background] Milano F, Gooley T, Wood B, Woolfrey A, Flowers ME, Doney K, Witherspoon R, Mielcarek M, Deeg JH, Sorror M, Dahlberg A, Sandmaier BM, Salit R, Petersdorf E, Appelbaum FR, Delaney C. Cord-Blood Transplantation in Patients with Minimal Residual Disease. N Engl J Med. 2016 Sep 8;375(10):944-53. doi: 10.1056/NEJMoa1602074. PMID 27602666
- [Background] Hiwarkar P, Qasim W, Ricciardelli I, Gilmour K, Quezada S, Saudemont A, Amrolia P, Veys P. Cord blood T cells mediate enhanced antitumor effects compared with adult peripheral blood T cells. Blood. 2015 Dec 24;126(26):2882-91. doi: 10.1182/blood-2015-06-654780. Epub 2015 Oct 8. PMID 26450984
- [Background] Admiraal R, Chiesa R, Lindemans CA, Nierkens S, Bierings MB, Versluijs AB, Hiwarkar P, Furtado Silva JM, Veys P, Boelens JJ. Leukemia-free survival in myeloid leukemia, but not in lymphoid leukemia, is predicted by early CD4+ reconstitution following unrelated cord blood transplantation in children: a multicenter retrospective cohort analysis. Bone Marrow Transplant. 2016 Oct;51(10):1376-1378. doi: 10.1038/bmt.2016.116. Epub 2016 May 9. No abstract available. PMID 27159172
- [Background] Chiesa R, Gilmour K, Qasim W, Adams S, Worth AJ, Zhan H, Montiel-Equihua CA, Derniame S, Cale C, Rao K, Hiwarkar P, Hough R, Saudemont A, Fahrenkrog CS, Goulden N, Amrolia PJ, Veys P. Omission of in vivo T-cell depletion promotes rapid expansion of naive CD4+ cord blood lymphocytes and restores adaptive immunity within 2 months after unrelated cord blood transplant. Br J Haematol. 2012 Mar;156(5):656-66. doi: 10.1111/j.1365-2141.2011.08994.x. Epub 2012 Jan 9. PMID 22224700
- [Background] Politikos I, Lavery JA, Hilden P, Cho C, Borrill T, Maloy MA, Giralt SA, van den Brink MRM, Perales MA, Barker JN. Robust CD4+ T-cell recovery in adults transplanted with cord blood and no antithymocyte globulin. Blood Adv. 2020 Jan 14;4(1):191-202. doi: 10.1182/bloodadvances.2019000836. PMID 31935291
- [Background] Estcourt LJ, Stanworth SJ, Hopewell S, Doree C, Trivella M, Massey E. Granulocyte transfusions for treating infections in people with neutropenia or neutrophil dysfunction. Cochrane Database Syst Rev. 2016 Apr 29;4(4):CD005339. doi: 10.1002/14651858.CD005339.pub2. PMID 27128488
- [Background] Massey E, Harding K, Kahan BC, Llewelyn C, Wynn R, Moppett J, Robinson SP, Green A, Lucas G, Sadani D, Liakopoulou E, Bolton-Maggs P, Marks DI, Stanworth S. The granulocytes in neutropenia 1 (GIN 1) study: a safety study of granulocytes collected from whole blood and stored in additive solution and plasma. Transfus Med. 2012 Aug;22(4):277-84. doi: 10.1111/j.1365-3148.2012.01152.x. Epub 2012 May 16. PMID 22591484
- [Background] Hiwarkar P, Adams S, Gilmour K, Nataraj R, Bonney D, Poulton K, Wynn R. Cord blood CD8+ T-cell expansion following granulocyte transfusions eradicates refractory leukemia. Blood Adv. 2020 Sep 8;4(17):4165-4174. doi: 10.1182/bloodadvances.2020001737. PMID 32886752
- [Background] Bashir S, Stanworth S, Massey E, Goddard F, Cardigan R. Neutrophil function is preserved in a pooled granulocyte component prepared from whole blood donations. Br J Haematol. 2008 Mar;140(6):701-11. doi: 10.1111/j.1365-2141.2008.06996.x. PMID 18302716
- [Derived] Borrill R, Poulton K, Kusyk L, Routledge A, Bonney D, Hanasoge-Nataraj R, Powys M, Mustafa O, Campbell H, Senthil S, Dillon R, Jovanovic J, Morton S, James B, Rao K, Stanworth S, Konkel J, Wynn R. Granulocyte transfusion during cord blood transplant for relapsed, refractory AML is associated with massive CD8+ T-cell expansion, significant cytokine release syndrome and induction of disease remission. Br J Haematol. 2023 Aug;202(3):589-598. doi: 10.1111/bjh.18863. Epub 2023 May 21. PMID 37211883